CLINICAL TRIAL: NCT04862936
Title: The Analysis of Prediction Model of Elderly Patients Visiting Emergency Department in Taiwan Triage and Acuity Scale
Brief Title: The Prediction Model of Elderly Patients in Taiwan Triage and Acuity Scale
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Changhua Christian Hospital (Other); Taipei City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 202000012B0C502
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-01

CONDITIONS: Frail Elderly Syndrome; Triage
Keywords: Triage; Frailty; Geriatric
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the year of 2010, the Taiwan Ministry of Health and Welfare had implemented the 5-level Taiwan Triage and Acuity Scale(TTAS) in Taiwan emergency department. TTAS is a triage system that was modified from CTAS. It has a comprehensive chief complaint system and accomplished with an electronic decision support system (eTTAS) to help triage nurse to assign acuity level on emergency patients in emergency departments of Taiwan. TTAS has adult and children modifiers, but no modifier for the elderly. In emergency departments, the geriatric population have been increasing in many countries for the last few years. They often present with atypical symptoms or signs, and multiple comorbidities that complicate diagnosis and treatment and are at risk of under-triage. Although the TTAS has overall validity and reliability, its performance in geriatric patients has not been well studied.

In order to reduce the chance to under-triage the geriatric patients in emergency departments and to improve the discriminatory and predictive power for triaged patients who require admission, the objective of the study is to examine the difference of urgency, admission rate and medical resource consumption of geriatric patients with different age group compared to non-geriatric patients, to develop predictive model for hospitalization and medical resource consumption among geriatric patients and to develop special geriatric modifiers.

DETAILED DESCRIPTION:
Age and frailty have been demonstrated to be associated with clinical outcomes in the elderly presented to emergent departments (EDs). This study aimed to assess the association of age and frailty on admission rate and to find out whether the current Taiwan Triage and Acuity Scale (TTAS) under-triage elderly presented to EDs.

This was a retrospective cohort study that reviewed medical records of adult patients from a single ED from 2016 to 2017. Data collected included patients' demographics, TTAS level, chief complaints, frailty status, and intensive care unit (ICU) admission rate. Adults patients included in the study were divided into three age groups of 18-<65, 65-85, and >85 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years old who go to the emergency department.
* Those who are willing to participate in the trial and sign a consent form and are willing to be tracked.

Exclusion Criteria:

* Patients under 65 years old who go to the emergency department.
* Patients over 65 years old who go to the emergency department, unwilling to participate in the trial and sign the consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 65 years old who go to the emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
admission rate | 1 day (since patient come into ER until he leave from ER.)
frailty scale | 1 day (since patient come into ER until he leave from ER.)

CONTACTS AND LOCATIONS:
Overall Officials: Chip Jin Ng, Dr., Principal Investigator — Chang Gung Memorial Hospital; Tsung Hsien Chao, Dr., Study Director — Chang Gung Memorial Hospital; Cheng Yu Chien, Dr., Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the first author on reasonable request.including
Supporting Information: Study Protocol, SAP, CSR, Analytic Code